CLINICAL TRIAL: NCT01235715
Title: The Use of Evicel to Reduce Blood Loss in Total Knee Replacement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 29054
Record Dates: First submitted 2010-10-08; First posted 2010-11-05 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-08

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; total knee replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evicel (Active Comparator): Evicel is a fibrin sealant used for hemostasis when control of bleeding by ligature or other conventional procedures is ineffective or impractical. It has been shown to stop bleeding in 2 minutes or less. Evicel is a combination of a biologic activated component containing human fibrinogen and topical thrombin that functions on wet, actively bleeding tissue. It is a bioresorbable and biocompatible agent.
  Interventions: Drug: Evicel fibrin sealant
- no evicel (No Intervention): Patients will receive standard treatment for bleeding as practiced at the Hospital for Special Surgery.

INTERVENTIONS:
Drug: Evicel fibrin sealant — Used for hemostasis to control bleeding. It has been shown to stop bleeding in 2 minutes or less. It is a combination of a biologic activated component containing human fibrinogen and topical thrombin functioning on wet, actively bleeding tissue.
  Arms: Evicel

SUMMARY:
Application of "Evicel" hemostatic matrix during operation for unilateral total knee replacement surgery (TKA) will result in decreased bleeding and postoperative drain output, a reduction in transfusion requirements, and less reduction of hemoglobin.

DETAILED DESCRIPTION:
No additional data desired

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of degenerative joint disease of the knee in patients medically suitable to undergo unilateral total knee arthroplasty

Exclusion Criteria:

* Known allergies to human blood products.
* History of bleeding disorders.
* Patients with previous arthrotomy, however, with exception of medial or lateral menisectomy.
* Patients taking Lovenox, Plavix, Aggrenox or erythropoetin. (coumadin is acceptable)
* Additionally, any patient with an intra-operative complication (i.e bone fracture, vascular injury) or post-operative complication that would affect bleeding tendency will be excluded although data will be recorded for later analysis. Also, any patient who has a complication with the suction drain (eg inadvertently being pulled out, suction failing) will have the remaining data points recorded and drain measurements will be excluded from analysis.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Figgie, M.D, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- See also: Ethicon website — http://www.ethicon360.com/products/evicel-fibrin-sealant-human

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing total knee arthroplasty at the Hospital for Special Surgery from September 2010 to June 2012 were enrolled in a consecutive prospective manner on a voluntary basis.
Groups:
- No Evicel: Patients will receive standard treatment for bleeding as practiced at HSS.
Period: Overall Study
Arm/Group | Evicel | No Evicel
Started | 98 | 102
Completed | 98 | 100
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Evicel | no Evicel | Total
Number analyzed (Participants) | 98 | 102 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 41 | 75
  >=65 years | 64 | 61 | 125
Age Continuous [Mean (Standard Deviation); unit: years] | 68.12 (9.88) | 66.38 (8.47) | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 59 | 116
  Male | 41 | 43 | 84
Region of Enrollment [Number; unit: participants]
  United States | 98 | 102 | 200

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin on Day 0 Compared to Preoperatively
Time Frame: preoperatively and on the day of surgery
Population: All patients enrolled in study were subject to analysis; occasionally a patient's levels were not taken or were not available for analysis for various reasons.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Evicel | No Evicel
Number analyzed (Participants) | 95 | 96
g/dL | -1.548 (.745) | -1.458 (.815)

2. Secondary Outcome: Change in International Normalized Ratio (INR) Level on Day 2 Compared to Preoperatively
Description: The INR, a measure of the clotting tendency of blood, is a ratio of a patient's prothrombin time (the time a blood plasma takes to clot after the addition of tissue factor) to a normal prothrombin time.
Time Frame: preoperatively and two days after surgery
Population: All patients who completed the study were included in analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Evicel | No Evicel
Number analyzed (Participants) | 98 | 100
ratio | .363 (.421) | 0.309 (0.514)

3. Secondary Outcome: Range of Motion on Day 3
Description: A measurement of the degrees of motion of the operated knee three days after surgery.
Time Frame: 3 days postoperatively
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Evicel | no Evicel
Number analyzed (Participants) | 98 | 100
degrees | 112.4 (1.983) | 114.1 (1.983)

4. Secondary Outcome: Visual Analog Pain Scale on Day 3
Description: The visual analog pain scale is a patient-reported measure of pain on a 10-point scale with 0 being no pain and 10 being worst possible pain. Drawings of faces indicate the level of pain associated with different points on the scale.
Time Frame: 3 days postoperatively
Measure: Mean (Standard Error); unit: points on VAS scale
Arm/Group | Evicel | no Evicel
Number analyzed (Participants) | 98 | 100
points on VAS scale | 4.3 (1.983) | 3.9 (1.983)

5. Primary Outcome: Change in Hematocrit on Day 0 Compared to Preoperatively
Time Frame: preoperatively and day of surgery
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of red blood cell
Arm/Group | Evicel | No Evicel
Number analyzed (Participants) | 94 | 96
percentage of red blood cell | -4.639 (2.275) | -4.220 (2.537)

6. Primary Outcome: Change in Hemoglobin On Day 1 Compared to Preoperatively
Time Frame: preoperatively and one day after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Evicel | No Evicel
Number analyzed (Participants) | 95 | 99
g/dL | -2.607 (0.986) | -2.480 (1.063)

7. Primary Outcome: Change in Hematocrit on Day 1 Compared to Preoperatively
Time Frame: preoperatively and one day after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of red blood cell
Arm/Group | Evicel | No Evicel
Number analyzed (Participants) | 94 | 99
percentage of red blood cell | -7.382 (2.801) | -7.199 (3.381)

8. Primary Outcome: Change in Hemoglobin on Day 2 Compared to Preoperatively
Time Frame: preoperatively and two days after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Evicel | No Evicel
Number analyzed (Participants) | 94 | 98
g/dL | -3.419 (1.437) | -3.497 (1.157)

9. Primary Outcome: Change in Hematocrit on Day 2 Compared to Preoperatively
Time Frame: preoperatively and two days after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of red blood cell
Arm/Group | Evicel | No Evicel
Number analyzed (Participants) | 93 | 98
percentage of red blood cell | -9.676 (4.540) | -10.100 (3.597)

10. Primary Outcome: Drain Output
Description: A measurement of the amount of blood drained from the knee.
Time Frame: 24 hours post-operatively
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mL
Arm/Group | Evicel | no Evicel
Number analyzed (Participants) | 98 | 100
mL | 780 (54.23) | 673 (54.23)

11. Primary Outcome: Number of Autologous Transfusion Units Over the Course of the Hospital Stay
Description: Units of autologous transfusion for each patient over the course of the hospital stay (an average of 3 days) were recorded.
Time Frame: perioperatively
Measure: Mean (Standard Error); unit: units
Arm/Group | Evicel | no Evicel
Number analyzed (Participants) | 98 | 100
units | 0.38 (0.041) | 0.46 (0.041)

12. Primary Outcome: Units of Homologous Transfusion Over the Course of the Hospital Stay
Description: Units of homologous transfusion for each patient over the course of the hospital stay (an average of 3 days) were recorded.
Time Frame: three days postoperatively
Population: All patients who completed the study were included in analysis.
Measure: Median (Standard Deviation); unit: units
Arm/Group | Evicel | No Evicel
Number analyzed (Participants) | 98 | 100
units | 0.276 (0.729) | 0.228 (0.581)

13. Secondary Outcome: Range of Motion at 6 Weeks
Description: A measurement of the degrees of motion of the operated knee six weeks after surgery.
Time Frame: 6 weeks postoperatively
Population: Patients whose range of motion at 6-week followup appointment was taken were included in analysis.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Evicel | no Evicel
Number analyzed (Participants) | 96 | 98
degrees | 114 (10.8) | 115 (12.4)

14. Secondary Outcome: Visual Analog Pain Scale (at Rest) at 6 Weeks
Description: The visual analog pain scale is a patient-reported measure of pain on a 10-point scale with 0 being no pain and 10 being worst possible pain. Drawings of faces indicate the level of pain associated with different points on the scale. For the measure of pain at rest, the patient indicates their level of pain while seated or lying down, not moving.
Time Frame: 6 weeks postoperatively
Population: Patients whose visual analog pain scale at 6-week followup appointment was taken were included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Evicel | no Evicel
Number analyzed (Participants) | 95 | 100
units on a scale | 1.326 (1.362) | 1.615 (1.801)

15. Secondary Outcome: Visual Analog Pain Scale (During Activity) at 6 Weeks
Description: The visual analog pain scale is a patient-reported measure of pain on a 10-point scale with 0 being no pain and 10 being worst possible pain. Drawings of faces indicate the level of pain associated with different points on the scale. For the measure of pain during, the patient indicates their level of pain while doing activities of daily living such as walking and moving from sitting to standing.
Time Frame: 6 weeks postoperatively
Population: Patients whose visual analog pain scale at 6-week followup appointment was taken were included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Evicel | no Evicel
Number analyzed (Participants) | 95 | 100
units on a scale | 2.821 (1.972) | 3.25 (2.167)

16. Secondary Outcome: Visual Analog Pain Scale (During Therapy) at 6 Weeks
Description: The visual analog pain scale is a patient-reported measure of pain on a 10-point scale with 0 being no pain and 10 being worst possible pain. Drawings of faces indicate the level of pain associated with different points on the scale. For the measure of pain during, the patient indicates their level of pain during physical therapy.
Time Frame: 6 weeks postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Evicel | no Evicel
Number analyzed (Participants) | 95 | 100
units on a scale | 4.479 (2.389) | 4.62 (2.597)

17. Secondary Outcome: Visual Analog Pain Scale (At Night) At 6 Weeks
Description: The visual analog pain scale is a patient-reported measure of pain on a 10-point scale with 0 being no pain and 10 being worst possible pain. Drawings of faces indicate the level of pain associated with different points on the scale. For the measure of pain at night, the patient indicates their level of pain during or before sleep.
Time Frame: 6 weeks postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Evicel | No Evicel
Number analyzed (Participants) | 95 | 99
units on a scale | 2.898 (2.192) | 2.813 (2.340)

ADVERSE EVENTS:
Arm/Group | Evicel | no Evicel
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/102
Other Adverse Events (participants affected / at risk) | 28/98 | 17/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evicel (N=98) | no Evicel (N=102)
Wound Healing Problem (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
GI Related Problems (Gastrointestinal disorders) | 5 (5) | 4 (4)
Cardiac or Blood Pressure Issues (Cardiac disorders) | 12 (12) | 8 (8)
Urinary Tract Infections (Renal and urinary disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 4 (4) | 3 (3)
Confusion (General disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No